CLINICAL TRIAL: NCT00762580
Title: Features to Predict Success With Nonoperative Treatment of Patients With Rotator Cuff Tears
Acronym: MOON
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: University of Colorado, Denver (Other); Ohio State University (Other); University of Iowa (Other); University of California, San Francisco (Other); Arthrex, Inc. (Industry); Knoxville Orthopedic Clinic (Other); Washington University School of Medicine (Other); Sports Medicine and Shoulder Surgery Orthopedic Institute (Unknown); Hospital for Special Surgery, New York (Other)
Responsible Party: Principal Investigator, Rosemary A. Sanders, Research Coordinator, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 060109
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Rotator Cuff Tear
Keywords: rotator cuff; rehabilitation
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Prospective: Patients with full thickness rotator cuff tears being treated with physical therapy

SUMMARY:
The goal of this study is to find which patients will improve with the nonsurgical treatment of physical therapy for the treatment of rotator cuff tears.

DETAILED DESCRIPTION:
Rotator cuff tears are found in up to 40% of people over the age of 50 with the prevalence increasing with age. While most people remain asymptomatic, it is unknown why some develop symptoms. In symptomatic patients, surgical repair of a torn rotator cuff fails in 30-50% of patients, yet the majority of patients have a significant reduction pain despite failure of the repair. Nonoperative treatment has reported successful outcomes in 25-82% of patients yet it is not known which patient-related features predict success with nonoperative treatment. The general aim of this research effort is to identify patient features (historical information, physical examination findings, and MRI-based pathology) that would predict success (defined by reduction in visual analog pain scale, and patient satisfaction) with the nonoperative treatment of rotator cuff tears. The proposed study design is a prospective cohort study of patients with rotator cuff tears who will follow a standard physical therapy program derived from an evidence based medicine (EBM) systematic review of Level 1 and Level 2 studies.

Study the effect of historical information on predicting success (as determined by pain relief and patient satisfaction) of nonoperative treatment using the EBM based physical therapy program in treating patients with rotator cuff tears.

Study the effect of physical examination findings on predicting success of a nonoperative treatment using the EBM-based physical therapy program in treating patients with rotator cuff tears.

Study the effect of the severity of the rotator cuff pathology (using standardized magnetic resonance imaging protocols) on predicting success of nonoperative treatment for patients with rotator cuff tears using the EBM-based physical therapy program.

ELIGIBILITY:
Inclusion Criteria:

• Patients (18-100 years of age) with MRI findings of a full-thickness rotator cuff tear

Note: Criteria to obtain a shoulder MRI to evaluate for rotator cuff tear [Appendix D]:

1. Significant weakness (≥ 2 points per guidelines above.)
2. ADL pain or night pain >/= 7 on VAS
3. Significant impingement (per guidelines above) + with significant symptoms for ≥ 3 months.

Exclusion Criteria:

* Acute rotator cuff tears (generally due to a high velocity injury and symptoms of less than one month)
* Associated dislocations
* Associated fractures
* Systemic Rheumatologic disease, i.e. Rheumatoid Arthritis and Systemic Lupus Erythematosis
* Patients being treated for bilateral rotator cuff tears simultaneously
* Patients unable to complete the forms
* Pain from neck or scapula
* Previous shoulder surgery
* Glenohumeral arthritis (meets ≥ 1 of below criteria)

  * osteophytes >2mm on humeral head or glenoid
  * Joint space narrowing with sclerosis or cyst formation seen on true AP or axillary radiographs;
  * humeral head contacting acromion
* Adhesive capsulitis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults between the ages of 18-100 with full thickness rotator cuff tears.
Sampling Method: Non-Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Predict successful outcome with an evidence-based, non-operative treatment program by collecting VAS Pain Scale and SANE score. | One year

SECONDARY OUTCOMES:
Predict success of non-operative treatment outcomes with other patient related validated instruments (SF-12, ASES, WORC, Marx Activity Scale) | One Year

CONTACTS AND LOCATIONS:
Overall Officials: John E. Kuhn, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (9):
- United States (9):
  - University of California at San Francisco, San Francisco, California
  - Colorado University Sports Medicine, Boulder, Colorado
  - Universtiy Of Iowa, Iowa City, Iowa
  - Department of Orthopaedic Surgery, Washington Universtiy School of Medicine, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - Ohio State, Columbus, Ohio
  - Sports Medicine & Shoulder Surgery, Orthopedic Institute, Sioux Falls, South Dakota
  - Shoulder and Elbow Institute, Knoxville Orthopaedic Clinic, Knoxville, Tennessee
  - Vanderbilt Universtiy Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
De Identified data from this cohort is only available to members of the MOON Shoulder Consortium. The member must provide a description of the use of the data to the research coordinator. The data request is then presented to the MOON consortium. A unanimous agreement of the plan by the consortium must be received prior to receiving the data.

REFERENCES:
- [Background] Bartolozzi A, Andreychik D, Ahmad S. Determinants of outcome in the treatment of rotator cuff disease. Clin Orthop Relat Res. 1994 Nov;(308):90-7. PMID 7955708
- [Background] Bokor DJ, Hawkins RJ, Huckell GH, Angelo RL, Schickendantz MS. Results of nonoperative management of full-thickness tears of the rotator cuff. Clin Orthop Relat Res. 1993 Sep;(294):103-10. PMID 8358901
- [Background] Chard MD, Hazleman R, Hazleman BL, King RH, Reiss BB. Shoulder disorders in the elderly: a community survey. Arthritis Rheum. 1991 Jun;34(6):766-9. doi: 10.1002/art.1780340619. PMID 2053923
- [Background] Charlson M, Szatrowski TP, Peterson J, Gold J. Validation of a combined comorbidity index. J Clin Epidemiol. 1994 Nov;47(11):1245-51. doi: 10.1016/0895-4356(94)90129-5. PMID 7722560
- [Background] Djurasovic M, Marra G, Arroyo JS, Pollock RG, Flatow EL, Bigliani LU. Revision rotator cuff repair: factors influencing results. J Bone Joint Surg Am. 2001 Dec;83(12):1849-55. doi: 10.2106/00004623-200112000-00013. PMID 11741065
- [Background] Ejnisman B, Andreoli CV, Soares BG, Fallopa F, Peccin MS, Abdalla RJ, Cohen M. Interventions for tears of the rotator cuff in adults. Cochrane Database Syst Rev. 2004;(1):CD002758. doi: 10.1002/14651858.CD002758.pub2. PMID 14973989
- [Background] Feng S, Guo S, Nobuhara K, Hashimoto J, Mimori K. Prognostic indicators for outcome following rotator cuff tear repair. J Orthop Surg (Hong Kong). 2003 Dec;11(2):110-6. doi: 10.1177/230949900301100202. PMID 14676334
- [Background] Galatz LM, Ball CM, Teefey SA, Middleton WD, Yamaguchi K. The outcome and repair integrity of completely arthroscopically repaired large and massive rotator cuff tears. J Bone Joint Surg Am. 2004 Feb;86(2):219-24. doi: 10.2106/00004623-200402000-00002. PMID 14960664
- [Background] Gerber C, Fuchs B, Hodler J. The results of repair of massive tears of the rotator cuff. J Bone Joint Surg Am. 2000 Apr;82(4):505-15. doi: 10.2106/00004623-200004000-00006. PMID 10761941
- [Background] Habernek H, Schmid L, Frauenschuh E. Five year results of rotator cuff repair. Br J Sports Med. 1999 Dec;33(6):430-3. doi: 10.1136/bjsm.33.6.430. PMID 10597856
- [Background] Harryman DT 2nd, Mack LA, Wang KY, Jackins SE, Richardson ML, Matsen FA 3rd. Repairs of the rotator cuff. Correlation of functional results with integrity of the cuff. J Bone Joint Surg Am. 1991 Aug;73(7):982-9. PMID 1874784
- [Background] Hattrup SJ. Rotator cuff repair: relevance of patient age. J Shoulder Elbow Surg. 1995 Mar-Apr;4(2):95-100. doi: 10.1016/s1058-2746(05)80061-8. PMID 7600171
- [Background] Itoi E, Tabata S. Conservative treatment of rotator cuff tears. Clin Orthop Relat Res. 1992 Feb;(275):165-73. PMID 1735208
- [Background] Itoi E, Tabata S. Incomplete rotator cuff tears. Results of operative treatment. Clin Orthop Relat Res. 1992 Nov;(284):128-35. PMID 1395281
- [Background] Kim SH, Ha KI, Park JH, Kang JS, Oh SK, Oh I. Arthroscopic versus mini-open salvage repair of the rotator cuff tear: outcome analysis at 2 to 6 years' follow-up. Arthroscopy. 2003 Sep;19(7):746-54. doi: 10.1016/s0749-8063(03)00395-5. PMID 12966383
- [Background] Kirkley A, Griffin S, McLintock H, Ng L. The development and evaluation of a disease-specific quality of life measurement tool for shoulder instability. The Western Ontario Shoulder Instability Index (WOSI). Am J Sports Med. 1998 Nov-Dec;26(6):764-72. doi: 10.1177/03635465980260060501. PMID 9850776
- [Background] Knudsen HB, Gelineck J, Sojbjerg JO, Olsen BS, Johannsen HV, Sneppen O. Functional and magnetic resonance imaging evaluation after single-tendon rotator cuff reconstruction. J Shoulder Elbow Surg. 1999 May-Jun;8(3):242-6. doi: 10.1016/s1058-2746(99)90136-2. PMID 10389080
- [Background] Lehman C, Cuomo F, Kummer FJ, Zuckerman JD. The incidence of full thickness rotator cuff tears in a large cadaveric population. Bull Hosp Jt Dis. 1995;54(1):30-1. PMID 8541777
- [Background] Lopez JG, Ernst MD, Wright TW. Acromioplasty: comparison of outcome in patients with and without workers' compensation. J South Orthop Assoc. 2000 Winter;9(4):262-6. PMID 12141189
- [Background] Massoud SN, Levy O, Copeland SA. Subacromial decompression. Treatment for small- and medium-sized tears of the rotator cuff. J Bone Joint Surg Br. 2002 Sep;84(7):955-60. doi: 10.1302/0301-620x.84b7.12378. PMID 12358385
- [Background] Motycka T, Kriegleder B, Landsiedl F. Results of open repair of the rotator cuff--a long-term review of 79 shoulders. Arch Orthop Trauma Surg. 2001;121(3):148-51. doi: 10.1007/s004020000199. PMID 11262780
- [Background] Patel VR, Singh D, Calvert PT, Bayley JI. Arthroscopic subacromial decompression: results and factors affecting outcome. J Shoulder Elbow Surg. 1999 May-Jun;8(3):231-7. doi: 10.1016/s1058-2746(99)90134-9. PMID 10389078
- [Background] Romeo AA, Hang DW, Bach BR Jr, Shott S. Repair of full thickness rotator cuff tears. Gender, age, and other factors affecting outcome. Clin Orthop Relat Res. 1999 Oct;(367):243-55. PMID 10546622
- [Background] Sallay PI, Reed L. The measurement of normative American Shoulder and Elbow Surgeons scores. J Shoulder Elbow Surg. 2003 Nov-Dec;12(6):622-7. doi: 10.1016/s1058-2746(03)00209-x. PMID 14671531
- [Background] Sher JS, Uribe JW, Posada A, Murphy BJ, Zlatkin MB. Abnormal findings on magnetic resonance images of asymptomatic shoulders. J Bone Joint Surg Am. 1995 Jan;77(1):10-5. doi: 10.2106/00004623-199501000-00002. PMID 7822341
- [Background] Silverstein B, Welp E, Nelson N, Kalat J. Claims incidence of work-related disorders of the upper extremities: Washington state, 1987 through 1995. Am J Public Health. 1998 Dec;88(12):1827-33. doi: 10.2105/ajph.88.12.1827. PMID 9842381
- [Background] Silverstein B, Viikari-Juntura E, Kalat J. Use of a prevention index to identify industries at high risk for work-related musculoskeletal disorders of the neck, back, and upper extremity in Washington state, 1990-1998. Am J Ind Med. 2002 Mar;41(3):149-69. doi: 10.1002/ajim.10054. PMID 11920960
- [Background] Spangehl MJ, Hawkins RH, McCormack RG, Loomer RL. Arthroscopic versus open acromioplasty: a prospective, randomized, blinded study. J Shoulder Elbow Surg. 2002 Mar-Apr;11(2):101-7. doi: 10.1067/mse.2002.120915. PMID 11988719
- [Background] Tempelhof S, Rupp S, Seil R. Age-related prevalence of rotator cuff tears in asymptomatic shoulders. J Shoulder Elbow Surg. 1999 Jul-Aug;8(4):296-9. doi: 10.1016/s1058-2746(99)90148-9. PMID 10471998
- [Background] Thomazeau H, Boukobza E, Morcet N, Chaperon J, Langlais F. Prediction of rotator cuff repair results by magnetic resonance imaging. Clin Orthop Relat Res. 1997 Nov;(344):275-83. PMID 9372778
- [Background] Vitale MG, Krant JJ, Gelijns AC, Heitjan DF, Arons RR, Bigliani LU, Flatow EL. Geographic variations in the rates of operative procedures involving the shoulder, including total shoulder replacement, humeral head replacement, and rotator cuff repair. J Bone Joint Surg Am. 1999 Jun;81(6):763-72. doi: 10.2106/00004623-199906000-00003. PMID 10391541
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Worland RL, Arredondo J, Angles F, Lopez-Jimenez F. Repair of massive rotator cuff tears in patients older than 70 years. J Shoulder Elbow Surg. 1999 Jan-Feb;8(1):26-30. doi: 10.1016/s1058-2746(99)90050-2. PMID 10077792
- [Background] Worland RL, Lee D, Orozco CG, SozaRex F, Keenan J. Correlation of age, acromial morphology, and rotator cuff tear pathology diagnosed by ultrasound in asymptomatic patients. J South Orthop Assoc. 2003 Spring;12(1):23-6. PMID 12735621
- [Background] Yamaguchi K, Tetro AM, Blam O, Evanoff BA, Teefey SA, Middleton WD. Natural history of asymptomatic rotator cuff tears: a longitudinal analysis of asymptomatic tears detected sonographically. J Shoulder Elbow Surg. 2001 May-Jun;10(3):199-203. doi: 10.1067/mse.2001.113086. PMID 11408898
- [Background] Zanetti M, Jost B, Hodler J, Gerber C. MR imaging after rotator cuff repair: full-thickness defects and bursitis-like subacromial abnormalities in asymptomatic subjects. Skeletal Radiol. 2000 Jun;29(6):314-9. doi: 10.1007/s002560000203. PMID 10929412
- [Background] Ellman H, Kay SP, Wirth M. Arthroscopic treatment of full-thickness rotator cuff tears: 2- to 7-year follow-up study. Arthroscopy. 1993;9(2):195-200. doi: 10.1016/s0749-8063(05)80374-3. PMID 8461081
- [Background] Goutallier D, Postel JM, Gleyze P, Leguilloux P, Van Driessche S. Influence of cuff muscle fatty degeneration on anatomic and functional outcomes after simple suture of full-thickness tears. J Shoulder Elbow Surg. 2003 Nov-Dec;12(6):550-4. doi: 10.1016/s1058-2746(03)00211-8. PMID 14671517
- [Background] Hawker G, Melfi C, Paul J, Green R, Bombardier C. Comparison of a generic (SF-36) and a disease specific (WOMAC) (Western Ontario and McMaster Universities Osteoarthritis Index) instrument in the measurement of outcomes after knee replacement surgery. J Rheumatol. 1995 Jun;22(6):1193-6. PMID 7674255
- [Background] Irrgang JJ, Anderson AF. Development and validation of health-related quality of life measures for the knee. Clin Orthop Relat Res. 2002 Sep;(402):95-109. doi: 10.1097/00003086-200209000-00009. PMID 12218475
- [Background] McHorney CA, Ware JE Jr, Lu JF, Sherbourne CD. The MOS 36-item Short-Form Health Survey (SF-36): III. Tests of data quality, scaling assumptions, and reliability across diverse patient groups. Med Care. 1994 Jan;32(1):40-66. doi: 10.1097/00005650-199401000-00004. PMID 8277801
- [Background] Small NC, Sledge CB, Katz JN. A conceptual framework for outcomes research in arthroscopic meniscectomy: results of a nominal group process. Arthroscopy. 1994 Oct;10(5):486-92. doi: 10.1016/s0749-8063(05)80002-7. PMID 7999155
- [Background] Ciepiela MD, Burkhead WZ. Classification of Rotator Cuff Tears. In: Burkhead WZ, ed. Rotator Cuff Disorders.Lippincott Williams & Wilkins, 1996.
- [Background] Cohen J. A coefficient of agreement for nominal scales. Educational and Psychological Measurement 1960;20:37-46.
- [Background] Jost B, Pfirrmann CW, Gerber C, Switzerland Z. Clinical outcome after structural failure of rotator cuff repairs. J Bone Joint Surg Am. 2000 Mar;82(3):304-14. doi: 10.2106/00004623-200003000-00002. PMID 10724223
- [Background] McHorney CA, Ware JE Jr, Raczek AE. The MOS 36-Item Short-Form Health Survey (SF-36): II. Psychometric and clinical tests of validity in measuring physical and mental health constructs. Med Care. 1993 Mar;31(3):247-63. doi: 10.1097/00005650-199303000-00006. PMID 8450681
- [Background] Sonnabend DH, Watson EM. Structural factors affecting the outcome of rotator cuff repair. J Shoulder Elbow Surg. 2002 May-Jun;11(3):212-8. doi: 10.1067/mse.2002.122272. PMID 12070491
- [Background] Stewart AL, Hays RD, Ware JE Jr. The MOS short-form general health survey. Reliability and validity in a patient population. Med Care. 1988 Jul;26(7):724-35. doi: 10.1097/00005650-198807000-00007. No abstract available. PMID 3393032
- [Background] Wolfgang GL. Surgical repair of tears of the rotator cuff of the shoulder. Factors influencing the result. J Bone Joint Surg Am. 1974 Jan;56(1):14-26. No abstract available. PMID 4812158
- [Background] Iannotti JP, Bernot MP, Kuhlman JR, Kelley MJ, Williams GR. Postoperative assessment of shoulder function: a prospective study of full-thickness rotator cuff tears. J Shoulder Elbow Surg. 1996 Nov-Dec;5(6):449-57. doi: 10.1016/s1058-2746(96)80017-6. PMID 8981270
- [Background] Neer CS 2nd. Anterior acromioplasty for the chronic impingement syndrome in the shoulder: a preliminary report. J Bone Joint Surg Am. 1972 Jan;54(1):41-50. No abstract available. PMID 5054450